CLINICAL TRIAL: NCT05818683
Title: A Phase 1b Study of JNJ-78278343, a T-cell Redirecting Agent Targeting Human Kallikrein 2 (KLK2), in Combination With Either JNJ-63723283 (Cetrelimab), Taxane Chemotherapy, or Androgen Receptor Pathway Inhibitors for Metastatic Prostate Cancer
Brief Title: A Study of JNJ-78278343 in Combination With Either JNJ-63723283 (Cetrelimab), Taxane Chemotherapy, or Androgen Receptor Pathway Inhibitors for Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109321; 78278343PCR1003 (Other: Janssen Research & Development, LLC); 2022-503132-14-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Neoplasms; Metastatic Hormone-sensitive Prostate Cancer
MeSH Terms: interventions — cabazitaxel; Docetaxel; apalutamide; enzalutamide; darolutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-78278343 + Combination agent: Part 1 (Dose Escalation) and Part 2 (Dose Expansion) (Experimental): Participants will receive JNJ-78278343 and combination agent (cetrelimab, cabazitaxel, docetaxel, apalutamide, enzalutamide, Darolutamide, abiraterone acetate plus prednisone) during Part 1 (dose escalation). The dose of JNJ-78278343 will be escalated sequentially until a recommended phase 2 regimen (RP2R). Participants will receive JNJ-78278343 and combination agent treatment at the putative RP2R in Part 2 (dose expansion).
  Interventions: Drug: JNJ-78278343; Drug: Cetrelimab; Drug: Cabazitaxel; Drug: Docetaxel; Drug: Apalutamide; Drug: Enzalutamide; Drug: Darolutamide; Drug: Abiraterone acetate plus prednisone (AAP)

INTERVENTIONS:
Drug: JNJ-78278343 — JNJ-78278343 will be administered.
Drug: Cetrelimab — Cetrelimab will be administered by intravenous infusion.
  Other Names: JNJ-63723283
Drug: Cabazitaxel — Cabazitaxel will be administered by intravenous infusion.
Drug: Docetaxel — Docetaxel will be administered by intravenous infusion.
Drug: Apalutamide — Apalutamide will be administered orally.
Drug: Enzalutamide — Enzalutamide will be administered orally.
Drug: Darolutamide — Darolutamide will be administered orally.
Drug: Abiraterone acetate plus prednisone (AAP) — Abiraterone acetate plus prednisone (AAP) will be administered orally.

SUMMARY:
The purpose of this study is to identify the recommended phase 2 regimen(s) RP2R(s) of JNJ-78278343 and combination agent in Part 1 (dose escalation) and to determine safety at the putative RP2R(s) of JNJ-78278343 with the combination agent in Part 2 (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

* Part 1 A-G (all combination treatments) and Parts 2B-C (cabazitaxel, docetaxel): Metastatic castration-resistant prostate cancer (mCRPC) with confirmed adenocarcinoma of the prostate as defined by prostate cancer working group 3 (PCWG3); Parts 2D-G (apalutamide, enzalutamide, darolutamide, abiraterone acetate + prednisone [AAP]): mCRPC: Histologically confirmed adenocarcinoma of the prostate as defined by PCWG3, with a minimum PSA of 2 nanogram [ng]/milliliter (mL); Part 2H (apalutamide): (a) metastatic hormone-sensitive prostate cancer(mHSPC) with PSA greater than (>) 0.2 ng/mL despite being treated with next generation ARPI (apalutamide, enzalutamide, darolutamide) for between 180 and 365 days (inclusive); (b) Participant may not have progressed radiographically or have PSA progression while receiving androgen deprivation therapy (ADT) and ARPI, as defined by PCWG3
* Measurable or evaluable disease
* (a) Part 1A (cetrelimab) - Prior treatment for mCRPC with at least 1 prior androgen receptor pathway inhibitors (ARPI) (that is, abiraterone acetate, apalutamide, enzalutamide, darolutamide), or chemotherapy (example, docetaxel). (b) Part 1C and 2C (docetaxel), Part 1D (apalutamide), Part 1E and 2E (enzalutamide), Part 1F and 2F (darolutamide), and Part 1G and 2G (AAP)- Prior treatment with at least 1 prior ARPI (that is, apalutamide, enzalutamide, darolutamide, or abiraterone acetate). (C) Part 1B and 2B (cabazitaxel) - Prior treatment with at least 1 prior ARPI (ie, abiraterone acetate, apalutamide, enzalutamide, darolutamide) and docetaxel. (d) Part 2D (apalutamide) - Prior treatment with at least 1 prior ARPI (e) Part 2H (apalutamide)- Participant must not have received prior cytotoxic chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ functions

Exclusion Criteria:

* Active autoimmune disease within the 12 months prior to signing consent that requires systemic immunosuppressive medications
* Toxicity related to prior anticancer therapy that has not returned to Grade less than or equal to (<=) 1 or baseline levels (except for alopecia, vitiligo, Grade <=2 peripheral neuropathy)
* Solid organ or bone marrow transplantation
* Known allergies, or intolerance to any of the components (example, excipients) of JNJ-78278343, cetrelimab (Part 1A), cabazitaxel, Part 1B and 2B , docetaxel Part 1C and 2C , apalutamide (Part 1D and 2D and Part 2H), enzalutamide (Part 1E and 2E), darolutamide (Part 1F and 2F), or AAP (Part 1G and 2G)
* Significant infections or serious lung, heart or other medical conditions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity (DLT) | Up to 21 days after first dose of combination agent
  DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity or hematologic toxicity.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years 11 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome events, which will be graded by American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years 11 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better without evidence of bone progression according to Prostate Cancer Working Group 3 (PCWG3) criteria.
Prostate Specific Antigen (PSA) Response Rate | Up to 2 years 11 months
  PSA response rate is defined as the percentage of participants with a confirmed decline of PSA of 50 percent (%) or more from baseline.
Radiographic Progression-free Survival (rPFS) | Up to 2 years 11 months
  rPFS is defined time from the date of first dose of JNJ-78278343 until the date of objective disease progression or death, whichever comes first.
Time to Response (TTR) | Up to 2 years 11 months
  TTR is defined for the responders as the time from the date of first dose of to the date of first documented response that is subsequently confirmed.
Duration of Response (DOR) | Up to 2 years 11 months
  DOR is defined for participants who achieved response (PR or better) as the time between the date of initial documentation of response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3, or death due to any cause, whichever occurs first.
Part 2H: Composite Progression-Free Survival (PFS) | Up to 2 years 11 months
  Composite PFS is defined as time from start of treatment to the date of first occurrence of investigator determined disease progression (Response Evaluation Criteria in Solid Tumors [RECIST] or bone progression), pain, PSA progression, death or last disease assessment, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (15):
- United States (7):
  - Florida Cancer Specialists, Sarasota, Florida
  - Start Midwest, Grand Rapids, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Perlmutter Cancer Center at NYU Langone Brooklyn, Brooklyn, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Health, New York, New York
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
- Australia (4):
  - Icon Cancer Centre Kurralta Park, Kurralta Park
  - Macquarie University, Macquarie University
  - Peter MacCallum Cancer Centre, Melbourne
  - Princess Alexandra Hospital, Woolloongabba
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency